CLINICAL TRIAL: NCT00004022
Title: Immunotherapy for Malignant Melanoma - Phase II Trial of Autologous Cancer Antigen Specific Immunotherapy
Brief Title: Biological Therapy Following Surgery in Treating Patients With Stage III or Stage IV Melanoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Barbara Ann Karmanos Cancer Institute (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Purpose: Treatment
Other Study IDs: CDR0000067241; P30CA022453 (NIH); WSU-C-1403-ME; NCI-G99-1565
Record Dates: First submitted 1999-11-01; First posted 2004-09-13 (Estimated); Last update posted 2013-04-05 (Estimated); Status verified 2013-04

CONDITIONS: Melanoma (Skin)
Keywords: stage III melanoma; stage IV melanoma; recurrent melanoma
MeSH Terms: conditions — Melanoma | interventions — aldesleukin; FANG vaccine; Muromonab-CD3; Surgical Procedures, Operative

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Biological: aldesleukin
Biological: autologous tumor cell vaccine
Biological: muromonab-CD3
Biological: therapeutic autologous lymphocytes
Procedure: surgical procedure

SUMMARY:
RATIONALE: Biological therapies use different ways to stimulate the immune system and stop cancer cells from growing. Combining different types of biological therapies may kill more tumor cells.

PURPOSE: Phase II trial to study the effectiveness of biological therapy following surgery in treating patients who have stage III or stage IV melanoma.

DETAILED DESCRIPTION:
OBJECTIVES:

* Evaluate the efficacy of immunotherapy with irradiated autologous tumor cell vaccine and sargramostim (GM-CSF) followed by monoclonal antibody OKT3- activated T lymphocytes and interleukin-2 in combination with surgery in terms of response rate in patients with stage III or IV malignant melanoma.
* Determine the immunogenicity of malignant melanoma in this patient population.

OUTLINE: Patients are stratified according to extent of disease, extent of antigen specific response to vaccination, performance status (0 vs 1), prior therapy (yes vs no), and gender.

Patients undergo surgical resection of tumor on week 1. Within 1-2 weeks of surgery, patients are vaccinated with irradiated autologous tumor cells and sargramostim (GM-CSF), then receive GM-CSF alone intradermally at vaccination sites daily for 4 days. Patients are revaccinated 2 weeks later.

Patients undergo peripheral blood mononuclear cell collection two weeks after the second vaccination. Peripheral blood mononuclear cells are stimulated with anti-CD3 monoclonal antibody (OKT3) and interleukin-2, producing activated T lymphocytes. The activated T lymphocytes are infused IV over 1-6 hours followed by 5 doses of interleukin-2 IV every other day over 10 days. Treatment continues in the absence of disease progression or unacceptable toxicity.

Patients may receive one additional course of immunotherapy as above.

Patients are followed every 3 months for 2 years, then every 6 months thereafter.

PROJECTED ACCRUAL: A total of 60 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically proven stage III or IV malignant melanoma
* Resectable disease
* At least 50,000,000 viable cells obtained from surgical specimen for use in the immunization part of this study

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Performance status:

* SWOG 0 or 1

Life expectancy:

* At least 6 months

Hematopoietic:

* Granulocyte count at least 1,500/mm^3
* Platelet count at least lower limit of normal
* No active or recent uncontrolled bleeding

Hepatic:

* Bilirubin normal
* SGOT no greater than 2 times upper limit of normal (ULN) (no greater than 5 times ULN if liver metastases present)

Renal:

* Creatinine normal

Other:

* Negative stool guaiac
* No impaired immunity
* No uncontrolled diabetes
* No active uncontrolled infections
* No other serious disease
* No other malignancies within the past 5 years except curatively treated basal or squamous cell skin cancer or carcinoma in situ of the cervix

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* Not specified

Chemotherapy:

* No concurrent chemotherapy

Endocrine therapy:

* Not specified

Radiotherapy:

* Not specified

Surgery:

* See Disease Characteristics

Other:

* At least 2 weeks since prior therapy and recovered

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 1997-06; Primary Completion 2004-01 (Actual); Study Completion 2004-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Roy D. Baynes, MD, PhD, FACP, Study Chair — Barbara Ann Karmanos Cancer Institute
Locations (1):
- Barbara Ann Karmanos Cancer Institute, Detroit, Michigan, United States